## Statistical Analysis Plan (SAP)

Study No. MSK-002

A Randomized, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Amifampridine Phosphate in Subjects with MuSK Antibody Positive Myasthenia Gravis, and a Sample of AChR Antibody Positive Myasthenia Gravis Subjects

Version 1.0

**January 27, 2020** 

Prepared for Catalyst Pharmaceuticals, Inc. 355 Alhambra Circle, Suite 1250 Coral Gables, FL 33134

Prepared by
STATKING Clinical Services
759 Wessel Drive
Fairfield, OH 45014
513-858-2989

www.statkingclinical.com



**STATKING Clinical Services** 

## **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document. Approved by: 28 Jan 2020 Steven Miller, PhD **Chief Operating Officer and Chief Scientific Officer** Catalyst Pharmaceuticals, Inc. 355 Alhambra Circle, Suite 1250 Coral Gables, FL 33134 smiller@catalystpharma.com Authored by: Dennis Clason, PhD **Date Statistician STATKING Clinical Services** 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 313 dclason@statkingclinical.com Approved by (internal review): Lori Christman, PhD **Date** Statistician STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 317 lori@statkingclinical.com

## **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document. Approved by: Steven Miller, PhD Date **Chief Operating Officer and Chief Scientific Officer** Catalyst Pharmaceuticals, Inc. 355 Alhambra Circle, Suite 1250 Coral Gables, FL 33134 smiller@catalystpharma.com Authored by: Statistician STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 313 dclason@statkingclinical.com Approved by (internal review): Lori Christman, PhD Statistician STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 317

lori@statkingclinical.com

1-28-2020

Approved by:

Clare Geiger, RN

**Project Manager** 

STATKING Clinical Services

759 Wessel Drive

Fairfield, OH 45014

513-858-2989 ext. 304

clare@statkingclinical.com

## **Revision History**

This version (Version 1.0) is the first version of this Statistical Analysis Plan. However, on July 12, 2017, a draft version of this document was submitted to the FDA in sequence 0109 of IND 106,263 as part of a submission requesting review of a Special Protocol Assessment. The protocol (and indirectly the July 12, 2017 draft version of this SAP) was approved by the FDA on August 23, 2017. Subsequent to that, Catalyst evaluated the suitability of the proposed statistical methods and proposed revisions to them. Those proposed revisions are included in this document.

## **Table of Contents**

| 1.0 SYNOPSIS OF STUDY DESIGN PROCEDURES | 7 |
|------------------------------------------------------|----|
| 1.1 Design and Treatment | 7 |
| 1.2 Study Procedures | 7 |
| 1.3 Sample Size | 8 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 8 |
| 2.1 Types of Analyses | 8 |
| 2.2 Analysis Populations | 9 |
| 2.3 Missing Data Conventions | 9 |
| 2.4 Interim Analyses | 10 |
| 2.5 Study Center Considerations in the Data Analysis | 10 |
| 2.6 Documentation and Other Considerations | 10 |
| 3.0 ANALYSIS OF BASELINE SUBJECT CHARACTERISTICS | 10 |
| 4.0 ANALYSIS OF EFFICACY | 10 |
| 4.1 Description of Efficacy Variables | 11 |
| 4.2 Analysis of Efficacy Variables | 12 |
| 5.0 ANALYSIS OF SAFETY | 14 |
| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 15 |
| 6.1 Subject Completion | 15 |
| 6.2 Study Drug Administration and Compliance | 16 |
| 6.3 Subject Data Profiles | 16 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 17 |
| 8.0 REFERENCES | 20 |

| APPENDIX A – TABLES, FIGURES | AND LISTING SPECIFICATIONS | .21 |
|------------------------------|----------------------------|-----|
| APPENDIX B – TABLE SHELLS | | .23 |

## 1.0 Synopsis of Study Design Procedures

This study is a prospective, randomized, placebo-controlled, multicenter study to evaluate the efficacy and safety of amifampridine phosphate in subjects diagnosed with MuSK-MG and a sample of AChR-MG subjects. The objectives of this Phase 3 study are as follows:

## Primary:

- To characterize the overall safety and tolerability of amifampridine phosphate compared with placebo in subjects with MuSK-MG; and,
- To assess the clinical efficacy of amifampridine phosphate compared with placebo in subjects with MuSK-MG, based on change of the Myasthenia Gravis-Activities of Daily Living (MG-ADL) score from Day 0 (baseline).

## Secondary:

- To assess the clinical efficacy of amifampridine phosphate compared with placebo in subjects with MuSK-MG, based on change of the Quantitative Myasthenia Gravis (QMG) score from Day 0 (baseline); and,
- To assess the safety and qualitative change in MG-ADL and QMG efficacy assessments of amifampridine phosphate compared with placebo in a sample of subjects with AChR-MG.

## 1.1 Design and Treatment

Subjects will be randomized on Day 0 to either treatment group in a 1:1 ratio. The Investigational Product (IP) will be administered under double-blind conditions such that neither the Investigator nor subject knows if they are taking placebo or amifampridine phosphate.

Amifampridine phosphate (at the subject's optimal dose established prior to entering the randomization period of this trial) or placebo will be dispensed by the site pharmacist, according to the randomization schedule, to begin dosing after all Day 0 assessments are completed and continued for 11 days.

The amifampridine phosphate dose is 30 mg to 80 mg total daily dose (expressed in free base form), given in 3 to 4 divided doses, with no single dose > 20 mg.

## 1.2 Study Procedures

The planned duration of participation for each subject is 1 to 14 days for screening, followed by a roughly 4-week run-in period. The run-in period will consist of open-label amifampridine dose adjustments every 3-4 days to achieve at least a 2 point improvement in MG-ADL (an inclusion requirement), observed during a subject's visit to the clinic during week 3 of run-in, and dose titration to

the limit of tolerability and no higher than a maximum of 80 mg per day. The subject must be on a constant dose for a minimum of 7 days to be eligible for randomization. Eligible subjects will be randomly assigned to either amifampridine or placebo tablets in a blinded fashion for treatment over 11 days (Day 0 through Day 10) provided all inclusion and exclusion criteria are met. The treatment period will commence on the remainder of Day 0 and continue to Day 10. The following assessments will be performed at the beginning and end of the 11-day treatment period:

- Vital signs;
- Urine sample collection on Day 10 for evaluation of IP compliance by testing for amifampridine and its metabolite in the urine;
- · Complete Physical Examination;
- 12-lead Electrocardiogram (ECG);
- Myasthenia Gravis specific Activities of Daily Living (MG-ADL);
- Quantitative Myasthenia Gravis (QMG);
- Record concomitant medications;
- Monitor for adverse events (throughout the run-in and treatment periods).

#### 1.3 Sample Size

The study is powered with respect to the primary endpoint of change in MG-ADL score from baseline. The sample size of the study has approximately 60% power to detect a 2 point difference, a minimally clinically significant difference, in the mean change from baseline between amifampridine and placebo treatment groups with a total sample size of n=60, assuming a standard deviation of the MG-ADL scores of 3.5. The 60 subjects do not include the 10 AChR-MG subjects. AChR-MG subjects are not expected to be respond robustly and positively and therefore no attempt will be made to adequately power the study for this group of study subjects.

## 2.0 Data Analysis Considerations

## 2.1 Types of Analyses

Analyses will consist of summarizing efficacy and safety data. Unless otherwise stated, two-sided p-values <0.05 will be considered as statistically significant.

The following standards will be applied for the analyses unless otherwise specified. Simple summary descriptive statistics for continuous data are: n (number of non-missing observations), mean, median, standard deviation, minimum, and maximum. A frequency count and percentage will be used to summarize the categorical data. Summary statistics will be presented by treatment. All data collected will be presented in the by-subject data listings, sorted by subject and by time point, where appropriate.

## 2.2 Analysis Populations

The analysis populations are defined as follows:

**Safety:** The safety population will consist of all subjects who are enrolled in the study and have received at least one dose of study drug. (Subjects who begin the run-in period belong to the Safety Population whether they are randomized to a treatment or not.)

**Full Analysis Set, Intent to Treat Population [FAS (ITT)]:** This population consists of all randomized subjects who receive at least 1 dose of IP (amifampridine or placebo post randomization) and have at least one post-treatment efficacy assessment. Subjects will be compared for efficacy according to the treatment to which they were randomized, regardless of the treatment actually received.

**Per Protocol (PP):** This population is a subset of the FAS (ITT) population, excluding subjects with major protocol deviations. The PP population will include all subjects who:

- Have no major protocol deviations or inclusion/exclusion criteria deviations that might potentially affect the validity of the efficacy analysis, and
- Subjects who took at least 80% of the required treatment doses.

Subjects who discontinue with no post-randomization data (no Day 0 and no Day 10 data) will be excluded from all efficacy analyses but will be included in the safety analyses. Decisions on exclusion from the FAS (ITT) and PP Populations will be finalized before unblinding prior to database lock.

The FAS (ITT) population will be the primary data set for all effectiveness analyses. The Safety population will be used to analyze all safety variables and baseline characteristics. The PP population will be used for selected effectiveness analyses.

#### 2.2.1 Subgroup Definitions

Subgroup analyses for efficacy will be performed independently on the MuSK-MG and AChR-MG groups. No pooled analyses are planned.

#### 2.3 Missing Data Conventions

No missing value imputation will be used in this analysis. All analyses will be based on the observed data.

For subjects that discontinue prior to Day 10 due to treatment related disability ("Rescue"), the observations collected at the time of rescue will be analyzed with the other Day 10 observations. Evaluations obtained at the time of discontinuation will be included in the FAS (ITT) and PP analyses, as applicable.

## 2.4 Interim Analyses

There are no interim analyses planned for this study.

## 2.5 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI).

There will be no selective pooling (sub-grouping) of study centers in the analysis. All calculations will be made on the combined results of all centers.

#### 2.6 Documentation and Other Considerations

The data analyses will be conducted using SAS® Software, version 9.4 or later.

## 3.0 Analysis of Baseline Subject Characteristics

Baseline and demographic characteristics will be summarized by treatment and overall for all subjects in the safety population. Age and baseline height and weight will be displayed via summary statistics (mean, median, sample size, standard deviation, minimum, and maximum). Gender and ethnicity will be summarized via counts and percentages.

A detailed listing of demographics data for each subject will also be provided as shown in Appendix B.

## 4.0 Analysis of Efficacy

The primary and secondary efficacy analyses will be conducted on the FAS (ITT) and PP populations, with the FAS (ITT) population serving as the primary efficacy analysis set for the primary and secondary efficacy variables. For the efficacy variables, change from baseline (CFB) will be computed as the post-treatment result (usually Day 10) minus the Baseline result (Day 0). The post-treatment result for subjects who discontinued treatment early is the CFB computed using the primary variable obtained at the time of dropout.

The analysis of efficacy will employ a closed testing procedure. Statistical significance in terms of the family-wise error rate for secondary endpoints will be

controlled at an alpha level of 0.05. Control will be accomplished based on a hierarchical closed testing procedure<sup>1,2</sup>. A secondary endpoint will be declared to have a statistically significant treatment effect if it and all previous endpoints in the hierarchy (including the primary) have reached statistical significance. The procedure stops at the first test that does not produce a two-sided p-value less than 0.05. The hierarchy of endpoint testing is MG-ADL (Primary), QMG (first secondary), MG-ADL Binary Response (second secondary), and QMG Binary Response (third secondary).

## 4.1 Description of Efficacy Variables

## 4.1.1 Primary Efficacy Variables

The primary efficacy variable for the study is the change in MG-ADL score from Day 0 (baseline) to Day 10 for MuSK-MG subjects treated with amifampridine and placebo.

The calculations and analyses are shown in Section 4.2.1.

## 4.1.2 Secondary Efficacy Variables

The secondary and exploratory efficacy variables are the following:

- The change in QMG score from Day 0 (baseline) to Day 10 for MuSK-MG subjects treated with amifampridine and placebo.
- A binary indicator (0 or 1) of response defined as a change of 2 or more in MG-ADL score from baseline to Day 10 for MuSK-MG subjects treated with amifampridine and placebo.
- A binary indicator (0 or 1) of response defined as a change of 3 or more in QMG score from baseline to Day 10 for MuSK-MG subjects treated with amifampridine and placebo.

The calculations and analyses pertaining to each of the above variables are shown in Section 4.2.2.

## 4.1.3 Exploratory Analysis of the Response of AChR-MG Subjects to Treatment

As described in Section 1.3, AChR-MG subjects are not expected to respond robustly and positively to the treatment with amifampridine. Those subjects showing an improvement of 2, or more, in MG-ADL from treatment with amifampridine during run-in will be enrolled, randomized, and qualitatively evaluated for the change from Day 0 (baseline) in the MG-ADL score and QMG. The endpoints for this evaluation are:

- Summary statistics by treatment for the MG-ADL score for Day 0, Day 10, and change from Day 0 (baseline).
- Summary statistics by treatment for the QMG score for Day 0, Day 10, and change from Day 0 (baseline).

## 4.2 Analysis of Efficacy Variables

## 4.2.1 Primary Efficacy Analysis

Summary statistics for the MG-ADL Day 0 assessment, MG-ADL Day 10 assessment, and the corresponding change from baseline for MG-ADL (CFB-MGADL) will be presented by treatment. The mean MG-ADL Total Score by time will be plotted by treatment and MG type.

The primary analysis of CFB-MGADL will be performed by fitting a fixed effects linear model to the data with CFB as the response. The model will include terms for treatment and MG-ADL at Baseline. The test comparing the least squares (LS) means will be conducted to evaluate the treatment effect:

H<sub>A,0</sub>: LSMeanCFB-MGADL(A) = LSMeanCFB-MGADL(P) vs.
H<sub>A,1</sub>: LSMeanCFB-MGADL(A) ≠ LSMeanCFB-MGADL(P),

where LSMeanCFB-MGADL(A) is the MG-ADL change from baseline LS mean of the amifampridine treatment group and LSMeanCFB-MGADL(P) is the MG-ADL change from baseline LS mean of the placebo treatment group.

A sensitivity analysis of the results of the test of the primary endpoint (MG-ADL CFB) score will be conducted using a nonparametric randomization test. The randomization test will repeat the fixed effects model analysis specified above after permutations of the treatment group assignments have been randomly performed. The procedure will be repeated a minimum of 1,000 times. If the observed test statistic is found to be in either the upper or lower 0.025 tail of the randomization p-value distribution, the null hypothesis of no treatment difference is rejected. A histogram of the p-values resulting from the 1000 permutation ANOVAs will be displayed together with the location of the p-value derived from the observed test statistic.

A data listing of the primary efficacy data will be constructed as shown in Appendix B.

## 4.2.2 Secondary Efficacy Analysis

Summary statistics for the Quantitative Myasthenia Gravis (QMG) Day 0 assessment, QMG Day 10 assessment, and the corresponding change from baseline (CFB-QMG) will be presented by treatment.

The secondary analysis of CFB-QMG will be performed by fitting a fixed effects linear model to the data with CFB-QMG as the response. The model will include terms for treatment and QMG at Baseline. The test comparing the least squares (LS) means will be conducted to evaluate the treatment effect:

H<sub>A,0</sub>: LSMeanCFB-QMG(A) = LSMeanCFB-QMG(P) vs.
H<sub>A,1</sub>: LSMeanCFB-QMG(A) ≠ LSMeanCFB-QMG(P),

where LSMeanCFB-QMG(A) is the QMG change from baseline LS mean of the amifampridine treatment group and LSMeanCFB-QMG(P) is the QMG change from baseline LS mean of the placebo treatment group.

A data listing of the QMG efficacy data will be constructed as shown in Appendix B.

## **MG-ADL Binary Response**

The number and proportion of MuSK-MG subjects with at least a 2 point change in MG-ADL score at Day 10 relative to Day 0 will be presented by treatment. The proportion for each treatment group will be computed with the number of subjects at Day 0 for each treatment group as the denominator, regardless of whether or not they completed the Day 10 assessment, and the number of subjects with at least a 2 point change in MG-ADL score at Day 10 as the numerator. A logistic regression model will be fitted to the binary variable indicating at least 2 points change in MG-ADL score as a function of the treatment assignment (Amifampridine or placebo) and the baseline MG-ADL score. The point estimate and 95% confidence interval on the point estimate will be displayed.

#### **QMG Binary Response**

The number and proportion of MuSK-MG subjects with at least a 3-point change in QMG score at Day 10 relative to Day 0 will be presented by treatment. The proportion for each treatment group will be computed with the number of subjects at Day 0 for each treatment group as the denominator, regardless of whether or not they completed the Day 10 assessment, and the number of subjects with at least a 3 point change in QMG score at Day 10 as the numerator. A logistic regression model will be fitted to the binary variable indicating at least 3 points change in QMG score as a function of treatment assignment (Amifampridine or placebo) and the baseline QMG score. The point estimate and 95% confidence interval on the point estimate will be displayed.

All secondary efficacy data will be listed as shown in Appendix B.

## 4.2.3 Exploratory Efficacy Analysis

As noted above, AChR-MG subjects are not expected to respond positively to amifampridine treatment. No inferential statistics are planned for this subgroup.

Summary statistics (n, mean, standard deviation, minimum, median and maximum) by treatment for the MG-ADL score for Day 0, Day 10, and change from Day 0 (baseline) will be presented.

Summary statistics (n, mean, standard deviation, minimum, median and maximum) by treatment for the QMG score for Day 0, Day 10, and change from Day 0 (baseline) will be presented.

All exploratory efficacy data will be listed as shown in Appendix B.

## 5.0 Analysis of Safety

The safety variables for this study are:

- Adverse events (AE)
- Vital signs (screening, Days 1 and 10)
- Physical examination (screening, Day 1, and Day 10 or termination from study)
- Electrocardiogram (ECG)
- Clinical laboratory results
- Concomitant medications

#### **Adverse Events**

All AEs will be observed for each subject from enrollment until termination from the study. Prior to analysis, all AEs will be coded using MedDRA. Based on these coded terms, treatment emergent AEs (TEAEs) will be summarized using system organ class and preferred term by treatment and overall for all subjects in the safety population. This analysis will be repeated for serious TEAEs (TESAEs).

TEAEs will also be summarized by severity and relationship to IP. An overall summary table will provide the highest relationship and maximum severity observed per subject, as well as the counts of subjects with at least one TESAE.

All AEs will be listed, regardless of whether or not they were treatment emergent.

#### Vital Signs

Summary statistics (mean, median, sample size, standard deviation, minimum, and maximum) will be computed on the raw and change from baseline values for each vital sign parameter by time point, for each treatment. The screening time

point will serve as baseline. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

## **Physical Exam**

A shift table of physical exam results will be created showing the shifts in results by parameter relative to the normal ranges. The number and percentage of subjects with the following shifts will be presented: normal/normal, normal/low, normal/high, low/low, low/normal, low/high, high/low, high/normal, and high/high. The physical exam data collected at screening, Day 0 and Day 10 (or termination from the study) will be listed.

## Electrocardiogram

A table containing descriptive statistics for QTc values measured at screening, Day 0 and Day 10 (or termination from the study) and CFB by treatment will be created. A shift table showing normal/normal, normal/abnormal, abnormal/normal and abnormal/abnormal shifts as counts and percentages for Days 0 and 10 will be created. The ECG data collected will be listed.

## **Clinical Laboratory Results**

Tables containing descriptive statistics for serum chemistry, hematology and urinalysis values measured at screening (pre-treatment level, the baseline value), Day 0 and Day 10 (or termination from the study) and Change From Screen Level (CFS) for both Day 0 and Day 10 by treatment will be created. In addition, a shift table will be constructed to show the shifts in laboratory results by parameter relative to the normal ranges. The number and percentage of subjects with the following shifts will be presented: normal/normal, normal/low, normal/high, low/low, low/normal, low/high, high/low, high/normal, and high/high.

#### **Concomitant Medications**

A table of the WHO-coded medications will be constructed by treatment group and overall with medications summarized by anatomical therapeutic chemical (ATC) level 4 term and preferred term. The number and percent of subjects on each drug will be summarized. A data listing for all concomitant medications will be provided.

## 6.0 Other Relevant Data Analyses/Summaries

## **6.1 Subject Completion**

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of the number of subjects withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The table

will include summary counts and percentages by treatment. A data listing of all subject completion and withdrawal data will also be constructed.

## 6.2 Study Drug Administration and Compliance

Duration of treatment administration will be computed per subject as:

Duration (in days) = (Date of last dose) – (Date of randomization) + 1

Duration will be summarized using descriptive statistics by treatment group.

Compliance will be computed per subject as:

Compliance = 100%\*(Number consumed)/(Number prescribed),

where number prescribed is defined as the duration times the number of tablets to have been taken daily. Compliance will be summarized using descriptive statistics by treatment group.

#### 6.3 Subject Data Profiles

A Subject Data Profile listing will be provided. It will contain demographic information, randomization information, all endpoint assessments and laboratory measurements. See Appendix B, Data Listing 19 for full details. Some variation in the appearance of this table is acceptable to accommodate unformatted SAS® output provided that all information is present.

## 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | | Shown in Appendix B |
|---|---|---|---|
| 1 | Subject Disposition (All subjects) | Х | X |
| 2 | Demographics and Baseline Data Summary Statistics – Continuous Variables (Safety Population) | Х | Х |
| 3 | Demographics and Baseline Data Summary Statistics – Categorical Variables (Safety Population) | Х | Х |
| 4 | Summary of Study Drug Administration and Compliance | Х | X |
| 5 | (Safety Population) MG-ADL Total Score Summary Statistics by Time Point | X | X |
| 6 | and MG Type (FAS Population) MG-ADL Total Score Summary Statistics by Time Point and MG Type (PP Population) | X | |
| 7 | MG-ADL CFB Analysis (FAS Population) | Х | X |
| 8 | MG-ADL CFB Analysis (PP Population) | Х | |
| 9 | MG-ADL CFB ANOVA Table (FAS Population) | Х | X |
| 10 | MG-ADL CFB ANOVA Table (PP Population) | Х | |
| 11 | QMG Total Score Summary Statistics by Time Point and MG Type (FAS Population) | X | Х |
| 12 | QMG Total Score Summary Statistics by Time Point and MG Type (PP Population) | Х | |
| 13 | QMG Total CFB Analysis (FAS Population) | Х | Х |
| 14 | QMG Total CFB Analysis (PP Population) | Х | |
| 15 | QMG Total CFB ANOVA Table (FAS Population) | Х | X |
| 16 | QMG Total CFB ANOVA Table (PP Population) | Х | |
| 17 | MG-ADL Sensitivity Analysis (FAS Population) | X | X |
| 18 | MG-ADL Sensitivity Analysis (PP Population) | X | |
| 19 | MG-ADL Score Shift of At Least 2 Points, MuSK MG Subjects (FAS Population) | X | X |
| 20 | MG-ADL Score Shift of At Least 2 Points, MuSK MG Subjects (PP Population) | Х | |
| 21 | QMG Score Shift of At Least 3 Points, MuSK MG<br>Subjects (FAS Population) | Х | Х |
| 22 | QMG Score Shift of At Least 3 Points, MuSK MG<br>Subjects (PP Population) | Х | |
| 23 | Number and Percent of Subjects with Treatment Emergent Adverse Events (Safety Population) | Х | Х |
| 24 | Summary of Treatment Emergent Adverse Events (Safety Population) | Х | Х |
| 25 | Number and Percent of Subjects with Serious Treatment Emergent Adverse Events (Safety Population) | х | Х |
| 26 | Number and Percent of Subjects with Treatment Emergent Adverse Events by Relationship to Treatment (Safety Population) | х | Х |
| 27 | Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade (Safety Population) | х | х |
| 28 | ECG Shift Summary Statistics by Treatment (Safety Population) | Х | Х |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in Appendix B |
|---|---|---|---|
| 29 | ECG QTc Interval Summary Statistics by Time Point and Treatment (Safety Population) | Х | X |
| 30 | Serum Chemistry Clinical Laboratory Summary Statistics by Time Point and Treatment (Safety Population) | Х | Х |
| 31 | Hematology Clinical Laboratory Summary Statistics by Time Point and Treatment (Safety Population) | Х | |
| 32 | Urinalysis Clinical Laboratory Summary Statistics by Time Point and Treatment (Safety Population) | Х | |
| 33 | Serum Chemistry Shift Table by Treatment (Safety Population) | Х | Х |
| 34 | Hematology Shift Table by Treatment (Safety Population) | Х | |
| 35 | Urinalysis Shift Table by Treatment (Safety Population) | Х | |
| 36 | Vital Sign Parameters Summary Statistics (Safety Population) | Х | Х |
| 37 | Vital Signs Shift Table by Treatment (Safety Population) | Х | Х |
| 38 | Number and Percent of Subjects Taking Concomitant Medications by ATC Level 3 and Preferred Term (Safety Population) | Х | Х |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in<br>Appendix B |
|---|---|---|---|
| Fig1 | Mean MG-ADL Total Score by Time Point and MG Type (FAS Population) | X | X |
| Fig2 | Mean MG-ADL Total Score by Time Point and MG Type (PP Population) | X | |
| Fig3 | Mean QMG Total Score by Time Point and MG Type (FAS Population) | X | |
| Fig4 | Mean QMG Total Score by Time Point and MG Type (PP Population) | X | |
| Fig5 | Randomization Test Histogram for MG-ADL Total Score (FAS Population) | X | Х |
| Fig6 | Randomization Test Histogram for MG-ADL Total Score (PP Population) | Х | |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in Appendix B |
|---|---|---|---|
| DL1 | Subject Disposition Data Listing | Х | X |
| DL2 | Protocol Deviations Data Listing | X | Х |
| DL3 | Demographics Data Listing | X | Х |
| DL4 | Subjects Excluded from FAS Population Data Listing | X | Х |
| DL5 | Subjects Excluded from PP Population Data Listing | X | Х |
| DL6 | Medical History Data Listing | X | Х |
| DL7 | Prior and Concomitant Medications Data Listing | X | Х |
| DL8 | Adverse Events Data Listing | X | X |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix B |
|---|---|---|---|
| DL9 | Physical Exam Data Listing | X | X |
| DL10 | Vital Signs Data Listing | X | X |
| DL11 | ECG Data Listing | X | X |
| DL12 | Study Drug Administration Data Listing | X | X |
| DL13 | Serum Chemistry Data Listing | X | X |
| DL14 | Hematology Data Listing | X | X |
| DL15 | Urinalysis Data Listing | X | X |
| DL16 | Amifampridine Level Data Listing | X | X |
| DL17 | MG-ADL Data Listing | X | X |
| DL18 | QMG Data Listing | X | Х |
| DL19 | Subject Data Profile | X | X |

## 8.0 References

- 1. Jennison, C; Turnbull, B.W.; "Group Sequential methods with Applications to Clinical Trials"; Chapman & Hall/CRC Press; 1999
- 2. Marcus, R.; Peritz, E.; Gabriel, K.R.; "On closed Testing Procedures with Special Reference to ordered Analysis of Variance"; Biometrica **63**, 655-660 (1976)

## Appendix A - Tables, Figures and Listing Specifications

#### Orientation

Tables, figures, and listings will be displayed in landscape with the exception of the Subject Data Profile Listing (DL19), which will be in portrait layout.

## **Margins**

Margins will be 1 inch on all sides. Table, figure, and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### Headers

The table number will be on the second line of the title area. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, one line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (Date)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

#### **Table Disclaimer**

The format of the mock tables shown in the appendix of this Statistical Analysis Plan (SAP) will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

## **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

## **Computation Values for Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (e.g., for a missing day value, the value displayed is in mmm-yyyy format). When date computations are necessary, the following table indicates the substitutions used in order to make those computations.

| Scenario | Value Used for Computations |
|---|---|
| Start date – Missing month and day values | January 1 of the indicated year |
| Start date – Missing day values | The first day of the indicated month |
| Stop date – Missing month and day values | December 31 of the indicated year |
| Stop date – Missing day values | The last day of the indicated month |

Appendix B - Table Shells

Page x of y

Table 1. Subject Disposition (All subjects)
Catalyst Pharmaceuticals, Inc. - MSK-002

| | | | ampridine<br>N=xx) | | lacebo<br>N=xx) | 70 | verall |
|---|---|---|---|---|---|---|---|
| Screen Failures | | | , | • | · | | XX |
| Enrolled | | | XX | | XX | | xx |
| Completed | | xx | (xxx%) | XX | (xxx%) | xx | (xxx%) |
| Withdrawn | | XX | (xxx%) | XX | (xxx%) | XX | (xxx%) |
| Reason for Withdrawal | Adverse Event Lost To Follow-Up Death Physician Decision Protocol Deviation Study Terminated by Sponsor Withdrawal by Subject Other | xx<br>xx<br>xx<br>xx<br>xx<br>xx | (xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%) | XX<br>XX<br>XX<br>XX<br>XX | (xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%) | xx<br>xx<br>xx<br>xx<br>xx | (xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%) |

The denominator for all percentages in the table is the number of enrolled subjects in the respective treatment group and overall.

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 2. Demographics and Baseline Data Summary Statistics - Continuous Variables Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Variable | Treatment Group | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|
| Age (years) | Amifampridine | XXX | xxx | xxx | xxx | xxx | xxx |
| iige (şealə) | Placebo | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |
| Baseline Weight (kg) | Amifampridine | XXX | xxx | xxx | xxx | xxx | xxx |
| | Placebo | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |
| Baseline Height (cm) | Amifampridine | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | XXX | XXX | XXX | XXX | XXX | XXX |
| | Overall | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 3. Demographics and Baseline Data Summary Statistics - Categorical Variables Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Demographics<br>Variable | Category | Amifampridine $(N=xxx)$ | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|
| Gender | Male<br>Female | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 4. Summary of Study Drug Administration and Compliance Catalyst Pharmaceuticals, Inc. - MSK-002

Safety Population (N=xxx)

| Myasthenia Gravis | | Statistic | Amifampridine<br>(N=xxx) | Placebo<br>(N=xxx) |
|---|---|---|---|---|
| MuSK | Duration (days) | n | XXX | XXX |
| | | Mean (Std Dev) | xxx (xxx) | xxx (xxx) |
| | | Median | XXX | XXX |
| | | Minimum, Maximum | xxx, xxx | XXX, XXX |
| | Compliance (%) | n | xxx | xxx |
| | | Mean (Std Dev) | xxx (xxx) | xxx (xxx) |
| | | Median | xxx | xxx |
| | | Minimum, Maximum | xxx, xxx | XXX, XXX |
| AChR | Duration (days) | n | xxx | XXX |
| | | Mean (Std Dev) | xxx (xxx) | xxx (xxx) |
| | | Median | xxx | xxx |
| | | Minimum, Maximum | xxx, xxx | xxx, xxx |
| | Compliance (%) | n | xxx | XXX |
| | | Mean (Std Dev) | xxx (xxx) | xxx (xxx) |
| | | Median | xxx | xxx |
| | | Minimum, Maximum | xxx, xxx | xxx, xxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 5. MG-ADL Total Score Summary Statistics by Time Point and MG type Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)

| Myasthenia Gravis | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Type | Treatment | Time Point <sup>a</sup> | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| MuSK | Amifampridine | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | (Baseline) | | | | | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Day 0 | RAW | xxx | xxx | XXX | xxx | xxx | xxx |
| | | (Baseline) | | | | | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| AChR | Amifampridine | Day 0 | RAW | xxx | xxx | XXX | xxx | xxx | XXX |
| | | (Baseline) | | | | | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Day 0 | RAW | xxx | XXX | XXX | XXX | xxx | xxx |
| | | (Baseline) | | | | | | | |
| | | Post-Baseline | RAW | XXX | XXX | XXX | XXX | XXX | xxx |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | xxx |

Source Program: xxxxxxx.sas

Source Listing: Data Listing 17

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 10, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

b RAW = observed data entered in the database; CFB = change from baseline = Value at time point - Baseline value. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

# Table 7. MG-ADL CFB Analysis Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)

| Statistic <sup>a</sup> | Amifampridine | Placebo |
|---|---|---|
| n | xxx | xxx |
| Least Squares (LS) Mean of Change from Baseline (CFB) | xxx | xxx |
| Between-Treatment Difference in LS Means | xxx | |
| 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| P-value for Between-Treatment Difference in LS Means | XXX | |

Source Program: xxxxxxx.sas Source Listing: Data Listing 17

<sup>&</sup>lt;sup>a</sup> CFB for MG-ADL total score was modeled as the response, with fixed effects terms for treatment and MG-ADL at Baseline. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

# Table 9. MG-ADL CFB ANOVA Table Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)

| Source | Degrees of<br>Freedom | Sum of<br>Squares | Mean Sum<br>of Squares | F Statistic | p-Value |
|---|---|---|---|---|---|
| Treatment | xxx | xxxxx | xxxxx | xxxx | xxxx |
| Baseline MG-ADL | xxx | xxxxx | xxxxx | xxxx | xxxx |
| Error | xxx | xxxxx | xxxxx | | |
| Total | xxx | XXXXX | | | |

Source Program: xxxxxxx.sas
Source Listing: Data Listing 17

<sup>&</sup>lt;sup>a</sup> CFB for MG-ADL total score was modeled as the response, with fixed effects terms for treatment and MG-ADL at Baseline. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 11. QMG Total Score Summary Statistics by Time Point and MG Type Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)

| Median |
|--------|
| xxx |
| XXX |
| XXX |
| xxx |
| XXX |
| XXX |
| XXX |
| XXX |
| XXX |
| xxx |
| XXX |
| XXX |
| - |

<sup>&</sup>lt;sup>a</sup> The post-treatment result will be the result obtained on Day 10, unless the subject discontinued treatment early, in which case the post-treatment result may be obtained at an earlier time point.

Source Program: xxxxxxx.sas Source Listing: Data Listing 18

b RAW = observed data entered in the database; CFB = change from baseline = Value at time point - Baseline value.

<sup>&</sup>lt;sup>c</sup> Observed significance level (p-value) for Wilcoxon-Mann-Whitney test of equality of change from baseline distributions. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

# Table 13. QMG Total CFB Analysis Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)

| Statistic <sup>a</sup> | Amifampridine | Placebo |
|---|---|---|
| n | XXX | xxx |
| Least Squares (LS) Mean of Change from Baseline (CFB) | XXX | xxx |
| Between-Treatment Difference in LS Means | xxx | |
| 95% CI for Between-Treatment Difference in LS Means | (xxx, xxx) | |
| P-value for Between-Treatment Difference in LS Means | XXX | |

xxxxxxx.sas

Source Listing: Data Listing 18

<sup>&</sup>lt;sup>a</sup> CFB for QMG total score was modeled as the response, with fixed effects terms for treatment and QMG at Baseline. Table Creation Date: (DD-MMM-YYYY)

Page x of y

# Table 15. QMG CFB ANOVA Table Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)

| Source | Degrees of<br>Freedom | Sum of<br>Squares | Mean Sum<br>of Squares | F Statistic | p-Value |
|---|---|---|---|---|---|
| Treatment | xxx | xxxxx | xxxxx | xxxx | xxxx |
| Baseline QMG | XXX | xxxxx | xxxxx | xxxx | xxxx |
| Error | xxx | xxxxx | xxxxx | | |
| Total | xxx | xxxxx | | | |

a CFB for QMG total score was modeled as the response, with fixed effects terms for treatment and QMG at Baseline.

Table Creation Date: (DD-MMM-YYYY)

xxxxxxx.sas

Source Listing: Data Listing 17

Page x of y

Table 17. MG-ADL Sensitivity Analysis
Catalyst Pharmaceuticals, Inc. - MSK-002
FAS Population (N=xxx)

Statistic<sup>a</sup> MG-ADL Score

XXX

P-value for Between-Treatment Difference in LS Means

<sup>a</sup> P-value based on conducting a randomization test by running the fixed effects linear model analysis on permuted treatment assignments. For each of the xxxx permutations, CFB was modeled as the response for each endpoint, with fixed effects terms for

treatment and score at Baseline.
Table Creation Date: (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Source Listing: Data Listing 17, Data Listing 18

Page x of y

Table 19. MG-ADL Score Shift Of At Least 2 Points, MuSK MG Subjects
Catalyst Pharmaceuticals, Inc. - MSK-002
FAS Population (N=xxx)

| Treatment | Score change | | | | | | |
|---|---|---|---|---|---|---|---|
| | Less Than<br>2 points | 2 or more<br>Points | Total | Logistic<br>Regression<br>Parameter | Point<br>Estimate | 95% Confidence<br>Interval of<br>Estimate | p-valueª |
| Amifampridine<br>Conditional | xxx<br>(xx.x%) | xxx<br>(xx.x%) | xxx | Treatment<br>Baseline Score | xxxx<br>xxxx | (xxxx,xxxx)<br>(xxxx,xxxx) | xxxx<br>xxxx |
| Placebo<br>Conditional | xxx<br>(xx.x%) | xxx<br>(xx.x%) | xxx | | | | |
| Total | xxx<br>(xx.x%) | xxx<br>(xx.x%) | xxx | | | | |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas Source Listing: Data Listing 17

 $<sup>^{\</sup>text{a}}$  P-value for the test of the null hypothesis  $\beta$  = 0.
Page x of y

Table 21. QMG Score Shift Of At Least 3 Points, MuSK MG Subjects
Catalyst Pharmaceuticals, Inc. - MSK-002
FAS Population (N=xxx)

| | Score | change | _ | | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Less Than<br>3 points | 3 or more<br>Points | Total | Logistic<br>Regression<br>Parameter | Point<br>Estimate | 95%<br>Confidence<br>Interval of<br>Estimate | p-valueª |
| Amifampridine<br>Conditional | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx | Treatment<br>Baseline Score | xxxx | (xxxx, xxxx)<br>(xxxx, xxxx) | xxxx |
| Placebo<br>Conditional | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx | | | | |
| Total | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx | | | | |

Source Program: xxxxxxx.sas Source Listing: Data Listing 18

Table format will be repeated for the PP Population.

 $<sup>^{\</sup>rm a}$  P-value for the test of the null hypothesis  $\beta$  = 0. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 23. Number and Percent of Subjects with Treatment Emergent Adverse Events
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

| Adverse Event Category <sup>a</sup> : | Amifampridine (N=xxx) | Placebo (N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| Total Number of Treatment Emergent Adverse Events (TEAEs) | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%)<br>xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 24. Summary of Treatment Emergent Adverse Events
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxxx)

| | Amifampridine (N=xxx) | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Maximum TEAE Severity Grade | | | |
| Mild (Grade 1) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Moderate (Grade 2) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Severe (Grade 3) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Life-threatening (Grade 4) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Death (Grade 5) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Treatment | | | |
| Not Related | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One Serious TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 25. Number and Percent of Subjects with Serious Treatment Emergent Adverse Events
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

| Adverse Event Categorya: | Amifampridine<br>(N=xxx) | Placebo<br>(N=xxx) | Overall<br>(N=xxx) |
|---|---|---|---|
| Total Number of Serious TEAEs | xxx | xxx | xxx |
| Subjects with at Least One Serious TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 26. Number and Percent of Subjects with Treatment Emergent Adverse Events by Relationship to Treatment

Catalyst Pharmaceuticals, Inc. - MSK-002

Safety Population (N=xxx)

| | | Amifampridine<br>(N=xxx) | | | | Placebo<br>(N=xxx) |
|---|---|---|---|---|---|---|
| Adverse Event Categorya: | Not Related | Possibly | Probably | Not Related | Possibly | Probably |
| Total Number of TEAEs | xxx | xxx | xxx | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version XXX STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 27. Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

Part 1 of 2

### Amifampridine (N=xxx)

| Grade 1 | | rade 2 | Gra | ade 3 | Grade 4 | | Grade 5 | |
|---|---|---|---|---|---|---|---|---|
| xxx | | XXX | : | xxx | | xxx | | xxx |
| xxx (xxx | :%) xxx | (xxx%) | xxx | (xxx%) | XXX | (xxx%) | xxx | (xxx%) |
| xxx (xxx | .%) xxx | (xxx%) | xxx | (xxx%) | XXX | (xxx%) | XXX | (xxx%) |
| xxx (xxx | .%) xxx | (xxx%) | XXX | (xxx%) | xxx | (xxx%) | XXX | (xxx%) |
| XXX (XXX | (%) XXX | (xxx%) | XXX | (xxx%) | XXX | (xxx%) | XXX | (xxx%) |
| | xxx (xxx<br>xxx (xxx<br>xxx (xxx<br>xxx (xxx | xxx (xxx%) xxx xxx (xxx%) xxx xxx (xxx%) xxx xxx (xxx%) xxx xxx (xxx%) xxx xxx (xxx%) xxx xxx (xxx%) xxx xxx xxx (xxx%) xxx xx | xxx xxx xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx | xxx xxx xxx xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) | xxx xxx xxx xxx xxx (xxx%) xxx (xxx%) xxx | xxx xxx xxx xxx xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx (xxx%) | xxx xxx xxx xxx xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx xxx (xxx%) xxx (xxx%) xxx (xxx%) xxx |

STATKING Clinical Services (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

Table 27. Number and Percent of Subjects with Treatment Emergent Adverse Events by Severity Grade Catalyst Pharmaceuticals, Inc. - MSK-002

Safety Population (N=xxx)

Part 2 of 2

Placebo (N=xxx)

| | (N-XXX) | | |
|---|---|---|---|
| Adverse Event Category <sup>a</sup> : | Grade 1 | Grade 2 Grade 3 | Grade 4 Grade 5 |
| Total Number of TEAEs | xxx | xxx xxx | xxx xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) |
| System Organ Class 1<br>Preferred Term 1<br>Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) xxx (xxx%)<br>xxx (xxx%) xxx (xxx%)<br>xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) |
| System Organ Class 2<br>Preferred Term 1<br>Preferred Term 2 | xxx (xxx%)<br>xxx (xxx%) | xxx (xxx%) xxx (xxx%) | xxx (xxx%) xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

a Adverse events coded with MedDRA Coding Dictionary Version XXX.

Page x of y

## Table 28. ECG Shift Summary Statistics by Treatment Catalyst Pharmaceuticals, Inc. MSK-002 Safety Population (N=xxx)

| Treatment Groups | Day 0 (Baseline)<br>Normal/<br>End of Study <sup>a</sup> Normal | Day 0 (Baseline)<br>Normal/<br>End of Study <sup>a</sup> Abnormal | Day 0 (Baseline)<br>Abnormal/<br>End of Study <sup>a</sup> Normal | Day 0 (Baseline)<br>Normal/<br>End of Study <sup>a</sup> Abnormal |
|---|---|---|---|---|
| Amifampridine (N=xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Placebo (N=xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

<sup>&</sup>lt;sup>a</sup> End of study is Day 10 or day of withdrawal from study, whichever is earlier.

STATKING Clinical Services (month day, year)

Page x of y

Table 29. ECG QTc Interval Summary Statistics
By Time Point and Treatment
Catalyst Pharmaceuticals, Inc. MSK-002
Safety Population (N=xxx)

| Treatment | Visit | Data<br>Type <sup>a</sup> | n | Mean<br>(msec) | Std<br>Dev | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|
| Amifampridine | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | xxx | xxx |
| | Day 0 (Randomization) | RAW | xxx | xxx | xxx | xxx | XXX | Xxx |
| | | CFB | XXX | XXX | XXX | XXX | XXX | Xxx |
| | End of study | RAW | XXX | XXX | XXX | XXX | XXX | Xxx |
| | | CFB | XXX | XXX | XXX | xxx | XXX | XXX |
| Placebo | Screening (Baseline) | RAW | XXX | xxx | xxx | xxx | xxx | xxx |
| | Day 0 (Randomization) | RAW | XXX | XXX | xxx | xxx | XXX | Xxx |
| | | CFB | XXX | XXX | XXX | XXX | XXX | Xxx |
| | End of study | RAW | XXX | XXX | XXX | XXX | XXX | Xxx |
| | | CFB | XXX | xxx | XXX | XXX | XXX | xxx |

a CFB refers to Change From Baseline CFB = Value at time point - Screening value.

STATKING Clinical Services (month day, year)

Page x of y

Table 30. Serum Chemistry Clinical Laboratory Summary Statistics by Time Point and Treatment

Catalyst Pharmaceuticals, Inc. MSK-002

Safety Population (N=xxx)

Laboratory Panel: Serum Chemistry

| Parameter | Treatment | Visit | Data<br>Type <sup>a</sup> | n | Mean | Std<br>Dev | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|---|
| - | | | | | | | | | |
| xxxxxxxxxxxxxxxx | Amifampridine | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Randomization) | RAW | XXX | xxx | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | End of study | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Randomization) | RAW | xxx | xxx | XXX | xxx | XXX | XXX |
| | | Day 0 (Kandomizacion) | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | End of study | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Bha Or Seady | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | OLD | 212121 | 212121 | 212121 | 212121 | 717171 | 212121 |
| xxxxxxxxxxxxxxxx | Amifampridine | Screening (Baseline) | RAW | xxx | xxx | XXX | XXX | xxx | XXX |
| | - | 3 . | | | | | | | |
| | | Day 0 (Randomization) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | End of study | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | Placebo | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Randomization) | RAW | XXX | xxx | xxx | xxx | xxx | xxx |
| | | Day 0 (Randomizacion) | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | End of study | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Ena or scuay | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFD | AAA | AAA | AAA | AAA | AAA | AAA |

 $<sup>^{\</sup>mathrm{a}}$  CFB refers to Change From Baseline CFB = Value at time point - Screening value.

STATKING Clinical Services (month day, year)

Source Program: xxxxxxx.sas

Source Listing: Data Listing 13

The format of this table is repeated for hematology and urinalysis panels.

Page x of y

## Table 33. Serum Chemistry Shift Table by Treatment Catalyst Pharmaceuticals, Inc. MSK-002 Safety Population (N=xxx)

| | | | Baseline Low <sup>a</sup> | | | Baseline Normal | | | Baseline High | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | EoSb | EoS | EoS | EoS | EoS | EoS | EoS | EoS | EoS |
| Lab Parameter | Treatment | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| xxxxxxxxx | Amifampridine | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx (xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) |
| xxxxxxxx | Placebo | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | XXX<br>(%XX%) | xxx<br>(xxx%) | xxx<br>(xxx%) |

Source Program: xxxxxxx.sas Source Listing: Data Listing 13

#### Table repeats for hematology and urinalysis panels.

<sup>&</sup>lt;sup>a</sup> Shifts represent screening/end of study (EoS), where EoS is Day 10 or day of withdrawal from study, whichever is earlier. STATKING Clinical Services (month day, year)

Page x of y

Table 36. Vital Signs Parameters Summary Statistics
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

| | | | | | | | Std | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Vital Sign P | Parameter (units) | Visit | Data Type <sup>a</sup> | n | Mean | Dev | Min | Max | Median |
| - 15 11 | | | | | | | | | | |
| Amifampridine | xxxxxxxxx ( | (xxx) | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | End of Study <sup>b</sup> | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| Placebo | xxxxxxxxx ( | (xxx) | Screening (Baseline) | RAW | xxx | xxx | xxx | XXX | XXX | xxx |
| | | | Day 0 | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | End of Study <sup>b</sup> | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> CFB refers to Change From Baseline CFB = Value at time point - Screening value.

<sup>&</sup>lt;sup>b</sup> End of study is Day 10 or day of withdrawal from study, whichever is earlier.

Page x of y

## Table 37. Vital Signs Shift Table by Treatment Catalyst Pharmaceuticals, Inc. MSK-002 Safety Population (N=xxx)

| | | Baseline Low <sup>a</sup> | | | Ва | aseline Norm | al | Baseline High | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | · | EoS | EoS | EoS | EoS | EoS | EoS | EoS | EoS | EoS |
| Lab Parameter | Treatment | Low | Normal H | High | High Low | Normal | High | Low | Normal | High |
| xxxxxxxxx | Amifampridine | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxxx | Placebo | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx<br>(xxx%) | xxx (xxx%) |

STATKING Clinical Services (month day, year)

<sup>&</sup>lt;sup>a</sup> End of study (EoS) is Day 10 or day of withdrawal from study, whichever is earlier.

Page x of y

# Table 38. Number and Percent of Subjects Taking Concomitant Medications by ATC Level 3 and Preferred Term Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Concomitant Medication Category <sup>a,b</sup> | Amifampridine<br>(N=xxx) | Placebo<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|
| ATC Level 4 Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| ATC Level 4 Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |
| WHO Preferred Term | xxxx (xxxx%) | xxxx (xxxx%) | xxxx (xxxx%) |

a Concomitant medications coded with WHO Coding Dictionary xxxxxxxxxxxx.

b Concomitant medication categories will include anatomical therapeutic chemical (ATC) level 4 term followed by preferred term. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y





STATKING Clinical Services (DD-MMM-YYYY)

Figure format will be repeated for the PP Population and for Mean QMG Total Score.

Page x of y

Figure 5. Randomization Test Histogram for MG-ADL Total Score Catalyst Pharmaceuticals, Inc. - MSK-002 FAS Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY)

Figure format will be repeated for the PP Population.

Page x of y

Data Listing 1. Subject Disposition Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002

| | Subject | | | | |
|---|---|---|---|---|---|
| Treatment | No. | MG-Type | Disposition Status | Date of Disposition | Withdrawal Reason |
| XXXXXX | XXXX | xxxxxx | xxxxxxxxxxxxxxxxxx | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxx | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxx | XXXXXXXXXXXXXXXXXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 2. Protocol Deviations Data Listing
Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

| Treatment | Subject<br>No. | Date of<br>Deviation | Deviation Description | Deviation Major or<br>Minor |
|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxx |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 3. Demographics Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | | Informed | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | Consent | Date of | Age | | | Screening | |
| Treatment | No. | Date | Birth | (yrs) | Gender | Ethnicity | Weight (kg) | Height (cm) |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXXXXX | XXXXXX | XXXXXX | xxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 4. Subjects Excluded from FAS Population Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002
Safety Population (N=xxx)

| Treatment | Subject No. | Reason for Exclusion |
|-----------|-------------|--------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | xxxx | xxxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 5. Subjects Excluded from PP Population Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002

All Enrolled Subjects (N=xxx)

| Treatment | Subject No. | Reason for Exclusion |
|-----------|-------------|-------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 6. Medical History Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

MedDRA System Organ Classa/

| | Subject | MedDRA Preferred Term/ | | |
|---|---|---|---|---|
| Treatment | No. | CRF Verbatim Term | Start Date | Ongoing? |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXX |

<sup>&</sup>lt;sup>a</sup> Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 7. Prior and Concomitant Medications Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

WHO Preferred Terma/ Verbatim Drug Name/

| | | | Verbatim Drug Name/ | | | | |
|---|---|---|---|---|---|---|---|
| | | Subject | Indication/ | Start | Stop | | |
| _ | Treatment | No. | ATC Level 4 Term | Date | Date | Route | Ongoing? |
| | XXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | XXXXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxx | | | | |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxx | | | | |

a Concomitant medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 8. Adverse Events Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | | Start<br>Date and<br>Time/ | | MedDRA System<br>Organ Class <sup>a</sup> /<br>MedDRA Preferred | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | End Date | Treatment | Term/ | Severity | Relation to | | |
| Treatment | No. | and Time | Start Date | CRF Verbatim Term | Grade | Treatment | Serious? | Outcome |
| xxxxxx | xxxxxxxx | xxxxxx<br>xxxxxx/<br>xxxxxx<br>xxxxxx | xxxxxx<br>xxxxxx | ************************************** | xxxxxxx | xxxxxxx | xxx | xxxxxxx |
| xxxxxx | xxxxxxxx | xxxxxxx<br>xxxxxxx/<br>xxxxxxx<br>xxxxxxx | xxxxxx | ************************************** | xxxxxxx | xxxxxxx | xxx | xxxxxxx |

a Adverse events coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 9. Physical Exam Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | Subject | | Date | | | |
|---|---|---|---|---|---|---|
| Treatment | No. | Visit | Conducted | Body System | Result | Abnormality |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | | XXXXXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | | xxxxxxx | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxxx | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | xxxxxxxx | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 10. Vital Signs Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Treatment | Subject<br>No. | Visit | Date | Time | Temp. | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Heart<br>Rate<br>(bpm) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | xxx | xxx | xxx | xxx |
| | | | | xxxxx | XXX | xxx<br>xxx | xxx<br>xxx | xxx<br>xxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | xxx | xxx | xxx | xxx |
| | | | | XXXXX | xxx | xxx<br>xxx | xxx<br>xxx | XXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 11. ECG Data Listing Catalyst Pharmaceuticals - MSK-002 Safety Population (N=xxx)

| ECG Assessment/ If<br>Abnormal, Specify | QT<br>Interval | QRS<br>Duration | PR<br>Interval | Heart<br>Rate | Time | Date | Time Point | Age | MG Type | Subject<br>No. |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/ | xxxxx | XXXXX | xxxxx | XXXXX | xxxxx | xxxxx | Screen | xxxx | xxxx | xxxxxx |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | xxxxx | Day 0 | | | |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxx | xxxxx | XXXXX | xxxxx | xxxxx | xxxxx | Day 10 | | | |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 12. Study Drug Administration Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | | Treatment | | Treatment | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | Start | Treatment | Duration | Tablets | | Tablets | |
| Treatment | No. | Date | End Date | (Days) | Consumed | Dose (mg/day) | Prescribed <sup>a</sup> | Compliance (%)b |
| xxxxxx | XXXX | xxxxxx | xxxxxx | XXX | XXX | xxx | xxx | xxx |
| xxxxxx | xxxx | xxxxxx | xxxxxx | XXX | xxx | xxx | xxx | xxx |

<sup>&</sup>lt;sup>a</sup> Number of tablets prescribed is computed as the duration times the number of tablets to have been taken daily.

b Compliance is computed as 100%\*(number of tablets consumed)/(number of tables prescribed). STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 13. Serum Chemistry Data Listing Catalyst Pharmaceuticals - MSK-002 Safety Population (N=xxx)

| Assessment/ If Abnormal, | | Parameter | | | |
|---|---|---|---|---|---|
| Specify | Value | (Units) | Date | Time Point | Subject No. |
| xxxxxxx/ | XXXXX | XXXXX | XXXXX | XXXXXX | XXXXXX |
| xxxxxxxxxxxxxxx | | | | | |
| xxxxxxx/ | XXXXX | XXXXX | | | |
| XXXXXXXXXXXXXXXXX | | | | | |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 14. Hematology Data Listing Catalyst Pharmaceuticals - MSK-002 Safety Population (N=xxx)

| | | | Parameter | | Assessment/ If Abnormal, |
|---|---|---|---|---|---|
| Subject No. | Time Point | Date | (Units) | Value | Specify |
| XXXXXX | XXXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | xxxxxxxxxxxxxxx |
| | | | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | XXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 15. Urinalysis Laboratory Data Listing
Catalyst Pharmaceuticals - MSK-002
Safety Population (N=xxx)

| | | | Parameter | | Assessment/ If Abnormal, |
|---|---|---|---|---|---|
| Subject No. | Time Point | Date | (Units) | Value | Specify |
| XXXXXX | XXXXXX | XXXXX | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | xxxxxxxxxxxxxxx |
| | | | XXXXX | XXXXX | xxxxxxx/ |
| | | | | | XXXXXXXXXXXXXXXXX |

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 16. Amifampridine Levels Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | Subject | | Date of | Time of | Amifampridine Level |
|-----------|---------|----------|---------|---------|---------------------|
| Treatment | No. | Visit | Sample | Sample | (Units) |
| xxxxx | xxxx | xxxxxxx | xxxxxxx | xx:xx | ****** |
| xxxxxx | xxxx | xxxxxxxx | xxxxxxx | xx:xx | xxxxxxxxxxxxxxxxxx |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 17. MG-ADL Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | Subject | | Myasthenia Gravis | | Change from | Best-Case Imputed | Worst-Case |
|---|---|---|---|---|---|---|---|
| Treatment | No. | Visit | ADL Score | Baseline Value | Baseline | Value | Imputed Value |
| xxxxx | XXXX | xxxxxxx | xxxx | xxxx | xxxx | xxxx | xxxx |
| xxxxxx | xxxx | xxxxxxx | XXXX | xxxx | xxxx | xxxx | XXXX |

STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

#### Data Listing 18. QMG Data Listing Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| | Subject | | | |
|---|---|---|---|---|
| Treatment | No. | Visit | Item | Score |
| XXXXXX | XXXX | XXXXXXXX | Double Vision (Lateral Gaze) Sec. | XXXX |
| | | | Bothersome Ptosis (Upward Gaze) Sec. | xxxx |
| | | | Facial Muscles | xxxx |
| | | | Swallowing 4oz. Water (1/2 cup) | xxxx |
| | | | Speech Following Counting Aloud From 1-50 (Onset of Dysarthria) | xxxx |
| | | | Right Arm Outstretched (90°, sitting) Sec. | XXXX |
| | | | Left Arm Outstretched (90°, sitting) Sec. | XXXX |
| | | | Forced Vital Capacity | xxxx |
| | | | Right Hand Grip (kg) | xxxx |
| | | | Left Hand Grip (kg) | xxxx |
| | | | Head, Lifted (45%, supine) Sec. | xxxx |
| | | | Right Leg Outstretched (45-50%, supine) Sec. | xxxx |
| | | | Left Leg Outstretched (45-50%, supine) Sec. | xxxx |
| | | | TOTAL | xxxx |

Page 69 of 72

STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 19. Subject Data Profile Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Study Numbe | er: MSK-002 | Site: xxxxxxxxx | Subject ID: xxxxx | |
|---|---|---|---|---|
| Randomizati<br>Age (yrs): | on Code: xxxx | Treatment: xxxxxx Gender: xxxxxx | Dose: xxxxxx<br>Ethnicity: xxxxxxx | Dose Group: xxxx |
| Screening W | Weight (kg): xxxx | MG Type: xxxxxxxx | | |
| Endpoint Me | asurements | | | |
| Myasthenia | Gravis - Activities | of Daily Living Scores | | |
| Visit | Date | e | Score | CFB |
| Baseline | XX- | xxx-xxxxx Total | XXXXX | |
| Day x | XX- | xxx-xxxx Total | xxxxx | xxxxx |
| Ouantitativ | e Myasthenia Gravis | Scores | | |
| Visit | Date | Item | Score | CFB |
| Baseline | xx-xxx-xxxx | Double Vision Sec. | XXXXX | |
| | | Bothersome Ptosis | xxxxx | |
| | | Facial Muscles | XXXXX | |
| | | Swallowing | xxxxx | |
| | | Speech Following Counting From 1-50 | XXXXX | |
| | | Right Arm Outstretched | xxxxx | |
| | | Left Arm Outstretched | XXXXX | |
| | | Forced Vital Capacity | xxxxx | |
| | | Right Hand Grip (kg) | xxxxx | |
| | | Left Hand Grip (kg) | xxxxx | |
| | | Head, Lifted | xxxxx | |
| | | Right Leg Outstretched | xxxxx | |
| | | Left Leg Outstretched | XXXXX | |
| | | Limb Total | xxxxx | |
| | | Total | XXXXX | |
| Day x | xx-xxx-xxxx | Double Vision Sec. | xxxxx | xxxxx |
| | | Bothersome Ptosis | XXXXX | XXXXX |
| | | Facial Muscles | XXXXX | XXXXX |
| | | Swallowing | XXXXX | XXXXX |
| | | Speech Following Counting From 1-50 | XXXXX | XXXXX |
| | | Right Arm Outstretched | XXXXX | XXXXX |
| | | Left Arm Outstretched | XXXXX | XXXXX |
| | | Forced Vital Capacity | XXXXX | XXXXX |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx.

Page x of y

Data Listing 19. Subject Data Profile Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Study Number: | MSK-002 | Site: xxxxxxxxx | Subject ID: | XXXXX | |
|---|---|---|---|---|---|
| Quantitative 1 | Myasthenia Gravis Sco | pres | | | |
| Visit | Date | Item | | Score | CFB |
| Day x | xx-xxx-xxxx | Right Hand Grip (kg) | | xxxxx | XXXXX |
| | | Left Hand Grip (kg) | | XXXXX | XXXXX |
| | | Head, Lifted | | XXXXX | XXXXX |
| | | Right Leg Outstretched | | XXXXX | XXXXX |
| | | Limb Total | | XXXXX | XXXXX |
| | | Total | | XXXXX | XXXXX |
| Safety Measur | ements | | | | |
| Laboratory Va | | Deventer (veite) | Result | Alamanana la Conittaniana | |
| Visit | Date | Parameter (units) | | Abnormal Criterion | |
| Baseline | xx-xxx-xxx | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| Day v | xx-xxx-xxxx | XXXXXXXXXXXXXXXXXX | XXXX<br>XXXX | | |
| Day x | **-***-*** | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | ************* | XXXX | | |
| | | *************************************** | AAAA | | |
| Electrocardio | _ | | | | |
| Visit | Date | Parameter (units) | Result | Abnormal Criterion | |
| Baseline | xx-xxx-xxxx | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| Day x | xx-xxx-xxxx | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | XXXXXXXXXXXXXXXXX | XXXX | | |
| | | xxxxxxxxxxxxxxx | xxxx | | |
| Vital Sign Va | lues | | | | |
| Visit | Date | Parameter (units) | Result | Abnormal Criterion | |
| Baseline | xx-xxx-xxxx | xxxxxxxxxxxxxxx | XXXX | · | |
| | | XXXXXXXXXXXXXXXXXX | XXXX | | |

<sup>&</sup>lt;sup>a</sup> Adverse events coded with MedDRA Coding Dictionary Version xxx.

Page x of y

Data Listing 19. Subject Data Profile Catalyst Pharmaceuticals, Inc. - MSK-002 Safety Population (N=xxx)

| Study Number: MS | K-002 | Site: xxxxxxx | XXX | Subject ID: 2 | xxxxx |
|---|---|---|---|---|---|
| Vital Sign Value | s | | | | |
| Visit | Date | Parameter (units | ) | Result | Abnormal Criterion |
| Day x | xx-xxx-xxxx | XXXXXXXXXXXXXX | XXXX | XXXX | |
| | | XXXXXXXXXXXXXXX | XXXX | XXXX | |
| | | XXXXXXXXXXXXXXX | XXXX | XXXX | |
| | | XXXXXXXXXXXXXXX | XXXX | XXXX | |
| Day x | XX-XXX-XXXX | XXXXXXXXXXXXXXX | XXXX | XXXX | |
| | | XXXXXXXXXXXXXXX | XXXX | XXXX | |
| | | XXXXXXXXXXXXXXX | XXXX | xxxx | |
| | | XXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxx | | |
| Adverse Events | | | | | |
| Preferred Term | Date | System Organ Cla | ss | Severity | Treatment Related? |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxxx | xxxxxx | xxxx | |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxxx | xxxxx | xxxx | xxxxxxxxxx |
| XXXXXXXXX | xx-xxx-xxxx | xxxxxxxxxxxxxx | xxxxx | xxxx | xxxxxxxxxx |
| XXXXXXXXX | XX-XXX-XXXX | XXXXXXXXXXXXXXXX | XXXXXX | XXXX | XXXXXXXXXX |
| Concomitant Medi | cations | | | | |
| Preferred Term | Dose (units, freq) | Start Date | Stop Date | | |
| XXXXXXX | xxxxx (xxxx, xxxx) | xx-xxx-xxx | xx-xxx-xxx | | |

Source Program: xxxxxxx.sas

Table repeats per subject beginning on a new page.

a Adverse events coded with MedDRA Coding Dictionary Version xxx.